CLINICAL TRIAL: NCT05444777
Title: The Effect of Low Dose Ketamine on Narcotic Consumption in Patients Undergoing Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Dr. Saima Rashid, Senior Instructor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2387-Ane-ERC-12
Record Dates: First submitted 2021-03-17; First posted 2022-07-06 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Cholelithiasis
MeSH Terms: conditions — Cholelithiasis | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine group (Group K) (Experimental): Group K was given ketamine @ 0.5mg/kg (prepared by dilution in 0.9% normal saline in 10 ml syringe) at the time of wound closure.
  Interventions: Drug: Ketamine Hydrochloride
- Saline group (Group S) (Other): Group S was given saline in 10 ml syringe
  Interventions: Drug: Ketamine Hydrochloride

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Ketamine was given prior to wound closure.
  Other Names: ketasol

SUMMARY:
This double-blinded randomized control trial aims to analyze the effect of low dose Ketamine on narcotic consumption, in patients undergoing Laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* all ASA 1 and 2 patients undergoing Laparoscopic Cholecystectomy electively.

Exclusion Criteria:

* Hepatic and renal disease and ASA 3 and 4 patients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2013-01-17 (Actual); Primary Completion 2013-11-30 (Actual); Study Completion 2013-11-30 (Actual)

PRIMARY OUTCOMES:
pain score using Visual Analogue scale, ranging from 0 (minimum) and 10 (maximum), 3 and below showing no pain and scores above 3 showing moderate to severe pain. | Baseline on arrival in the post anaesthesia care unit and then every fifteen minutes unto one hour
  Change in pain score using Visual Analogue Scale

SECONDARY OUTCOMES:
narcotic consumption in the post operative anaesthesia care unit | postoperatively, after arrival in the post anaesthesia care unit at every fifteen minutes unto one hour
  requirement of narcotic in the post anaesthesia care unit

IPD SHARING:
Plan to Share IPD: No